CLINICAL TRIAL: NCT04612283
Title: A Double Blind, Randomized, Parallel Group Study to Evaluate Efficacy and Safety of NGA-01 Gel Against Placebo in the Treatment of Osteoarthritis With Joint Pain
Brief Title: NGA-01 Gel for the Treatment of Osteoarthritis With Joint Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nutrin GmbH (Network)
Collaborators: Galaxa Pharma (Unknown); Mittal Global Clinical Trial Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NUTRIN004
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Arthritis Osteoarthritis
Keywords: osteoarthritis; pain
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Pain

STUDY DESIGN:
Intervention Model Description: double blind, randomized, parallel group study against placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NGA-01 gel (Active Comparator): A formulation with natural ingredients expected to be used for joint pain in Osteoarthritis
  Interventions: Other: NGA-01 gel
- Placebo gel (Placebo Comparator): Placebo gel with no active ingredient
  Interventions: Other: Placebo

INTERVENTIONS:
Other: NGA-01 gel — NGA-01 is a gel formulation with mostly herbal active ingredients
  Arms: NGA-01 gel
Other: Placebo — A Placebo with no active ingredients
  Arms: Placebo gel

SUMMARY:
Osteoarthritis is characterized by the breakdown of cartilage in joints. As cartilage deteriorates, the bones of the joint begin to run against one another, causing stiffness and pain, which often impairs movement. Osteoarthritis also can damage ligaments, menisci, and muscles. Bone or cartilage fragments may float in the joint space, causing irritation and pain. Bone spurs, or osteophytes, may also develop, causing additional pain and potentially damaging surrounding tissues. Around the world, an estimated 10%-15% of adults over 60 have some degree of osteoarthritis. It most commonly affects the joints in the knee, hands, feet, and spine, and is also relatively common in other joints such as the shoulder and hip joints. There are two types of osteoarthritis: primary and secondary. Primary osteoarthritis is a chronic degenerative disease that is related to, but not caused by, aging. As a person ages, the water content of their cartilage decreases, thus weakening it and making it less resilient and more susceptible to degradation. There are strong indications that genetic inheritance is a factor, as up to 60% of all OA cases are thought to result from genetic factors. The main symptoms are pain, loss of ability, and "joint stiffness after exercise or use." These symptoms are often aggravated by activity or rigorous exercise and relieved during rest, though the disease may eventually progress to the point where the patient even feels pain when resting, and some people report pain so intense that it wakes them up when they are sleeping. Osteoarthritis, at present, cannot be cured, and will likely get worse over time, but the symptoms can be controlled. Treatments vary widely, from alternative medicine, to lifestyle changes such as exercise and diet, to physical aids such as canes or braces, to medications such as acetaminophen, nonsteroidal anti-inflammatory drugs (NSAIDS), corticosteroids, and more. Osteoarthritis is the most common joint disease of human. Among the elderly knee osteoarthritis is leading cause of chronic disability in developed countries. Some people in India are unable to walk independently from bed and bath-room because of Osteoarthritis of the knee or hip joint. Osteoarthritis (OA) also known as degenerative arthritis or degenerative joint disease, is a group of mechanical abnormalities involving degradation of joints, including articular cartilage and subchondral bone. Symptoms may include joint pain, tenderness, stiffness, locking, and sometimes an effusion. A variety of causes viz. hereditary, developmental, metabolic, and mechanical may initiate processes leading to loss of cartilage. When bone surfaces are not well protected by cartilage, bone may get exposed and damaged. As a result of decreased movement secondary to pain, atrophy of regional muscles, and ligaments may become more lax.

The goal of treatment is to reduce or eliminate the signs and symptoms of Osteoarthritis. Mild to moderate disease is often treated with topical therapies. Sponsor has developed the NGA-01Gel containing the fixed dose combination of alcohol and water mixture, with active herbal ingredients, without preservatives and dyes. The Gel is easy to apply, and the cosmetic appearance is that of a white, milky gel, easily-spreadable that absorbs completely into the skin a few minutes after application and it is expected that the Gel will differentiate from marketed formulations by patient preference for the gel and gel.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having at least one or more sign and symptoms of Osteoarthritis like Pain in joints (at Knee, Hip, Ankle, Elbow and Shoulder), stiffness, difficulty in flexion and extension, crepitus, swelling etc for more than 3 months prior to the study.
* Pain score of at least 4 cm on a 10-cm linear visual analogue scale.
* Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events.
* Are willing to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural or artificial) for the duration of the study.
* Are willing to refrain from using any lotions, gel, balm, moisturizer, cleansers, cosmetics or creams, other than those issued as part of the study, on the treatment areas during the treatment period.
* If female of childbearing potential, must be willing to practice an acceptable form of birth control for the duration of the study.
* Are able to give written informed consent in a manner approved by the Institutional Ethics Committee and comply with the requirements of the study.
* Are willing to avoid participation in any other interventional clinical trial for the duration of this study.

Exclusion Criteria:

* Are pregnant, breast-feeding, or planning to become pregnant during the study.
* Patients with Rheumatoid Arthritis, Systemic Lupus Erythematosus, Psoriatic Arthritis, Gouty Arthritis.
* Complications of OA, like Pseudogout, Spontaneous osteonecrosis of the knee, Ruptured Baker cyst, Bursitis, Anserine bursitis (knee)interfere with the disease and treatment.
* Severe Stomach infection.
* Severely traumatised and/or very severe or mucosal inflammation
* Peritonsillar abscess
* Long term use (≥ 3 times per week within the last month or regular intake within the last 3 months before randomisation) of antiinflammatory drugs- Any long-acting or slow release analgesic intake including Non Steroidal Anti-Inflammatory Drugs (NSAIDs)within 24 hours before randomisation (e.g. piroxicam or naproxen)
* Any anti-inflammatory drugs intake by systemic route within 12 hours before randomization
* Any paracetamol intake within 6 hours before randomisation
* Any cold medication (decongestant, antihistamine, expectorant, antitussive) within 6 hours before randomisation
* Heavy smokers (>10 cigarettes/day)
* Have open sores or open lesions in the treatment area(s).
* Have any condition that, in the opinion of the investigator, would confound the safety and/or efficacy assessments of plaque Arthritis.
* Have participated in any interventional clinical trial in the previous 30 days.
* Have a known sensitivity to any of the constituents of the test product
* Have used, are using, or are planning to use immunosuppressive or immunomodulatory medication (i.e., biologics), including oral or parenteral corticosteroids.
* Have a history of alcohol or illegal drug/substance abuse, or suspected alcohol or illegal drug/substance abuse in the past 2 years.
* Plan to seek alternative treatment of any kind for their Arthritis, in the eligible treatment areas or otherwise, during the trial period.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Change in pain visual analog scale (VAS) scores (0-10) from baseline | Day 0 - Day 60
  Pain was recorded as per physician's analysis as per SOP, 0 as lowest and 10 as highest

SECONDARY OUTCOMES:
Change in WOMAC scores | Day 0 - Day 60
  Western Ontario and McMaster Universities Arthritis Index is used to determine severity of arthritis
Change in Numeric Pain Rating Scale (NPRS) score | Day 0 - Day 60
  Pain is measured as per regular NPRS scale
Change in Range of motion (ROM) | Day 0 - Day 60
  physical assessment by the doctor
Change in Physician's Global Assessment of Arthritis | Day 0 - Day 60
  The physicians analysed data is recorded
Change in Patient's Global Assessment of Arthritis | Day 0 - Day 60
  The customer questionnaire based data is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Moraya Multispeciality Hospital, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
This is a blinded gel trial with efficacy and safety data to be evaluated. Being a confidential formulation, we are not very sure and have no plans to share any data till date.